CLINICAL TRIAL: NCT01821144
Title: A School-based Education Programme to Reduce Salt Intake in Children and Their Families (School-EduSalt)
Brief Title: A School-based Education Programme to Reduce Salt Intake in Children and Their Families
Acronym: School-EduSalt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: The George Institute for Global Health, China (Other); Peking University (Other); Changzhi Medical College (Other)
Responsible Party: Principal Investigator, Feng J He, Senior Research Fellow, Queen Mary University of London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 008602 QM
Record Dates: First submitted 2013-03-21; First posted 2013-03-29 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Healthy Volunteer
Keywords: dietary salt; 24 hour urinary sodium; blood pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): No salt awareness education
  Interventions: Other: Control
- Salt reduction (Experimental): Salt reduction
  Interventions: Behavioral: Salt reduction

INTERVENTIONS:
Behavioral: Salt reduction — Salt reduction
  Arms: Salt reduction
Other: Control — No salt awareness education
  Arms: Control

SUMMARY:
The study is to test whether an education programme targeted at school children can lower salt intake in children and their families. In this study, the investigators will educate children on how to reduce salt intake, and the investigators will empower children by asking them to deliver the salt reduction message home to their families, particularly children need to persuade the person who does the cooking for the whole family to cut down on the amount of salt used during food preparations. The study will involve children aged about 11 years, and their parents and grandparents in Northern China.

ELIGIBILITY:
Children

Inclusion Criteria:

* All children in Grade 5 of primary schools (age about 11 years) are eligible for the study.

Exclusion Criteria:

* Children who do not have lunch or dinner at their own home will be excluded.

Adult family members:

Inclusion Criteria:

* For each participating child, we will recruit two adult family members. All adult family members who share the same meals with the child are eligible for the study.

Exclusion Criteria:

* If more than two adults in one family agree to take part in the study, we will select two of them (i.e. one male and one female) in the order of grandparents, parents, uncles and aunties.

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 832 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
24-h urinary sodium | 4.5 month
  Difference between the intervention and control group in the change in 24-h urinary sodium from baseline to the end of follow-up for children and for adults

SECONDARY OUTCOMES:
Blood pressure | 4.5 month
  Difference between the intervention and control group in the change in blood pressure from baseline to the end of follow-up for children and for adults.

CONTACTS AND LOCATIONS:
Overall Officials: Feng He, PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- Changzhi Medical College, Changzhi, Shanxi, China

REFERENCES:
- [Derived] Ma Y, Feng X, Ma J, He FJ, Wang H, Zhang J, Xie W, Wu T, Yin Y, Yuan J, MacGregor GA, Wu Y. Social support, social network and salt-reduction behaviours in children: a substudy of the School-EduSalt trial. BMJ Open. 2019 Jun 14;9(6):e028126. doi: 10.1136/bmjopen-2018-028126. PMID 31203245
- [Derived] Li X, Jan S, Yan LL, Hayes A, Chu Y, Wang H, Feng X, Niu W, He FJ, Ma J, Han Y, MacGregor GA, Wu Y. Cost and cost-effectiveness of a school-based education program to reduce salt intake in children and their families in China. PLoS One. 2017 Sep 13;12(9):e0183033. doi: 10.1371/journal.pone.0183033. eCollection 2017. PMID 28902880
- [Derived] He FJ, Ma Y, Feng X, Zhang W, Lin L, Guo X, Zhang J, Niu W, Wu Y, MacGregor GA. Effect of salt reduction on iodine status assessed by 24 hour urinary iodine excretion in children and their families in northern China: a substudy of a cluster randomised controlled trial. BMJ Open. 2016 Sep 26;6(9):e011168. doi: 10.1136/bmjopen-2016-011168. PMID 27670515
- [Derived] He FJ, Wu Y, Feng XX, Ma J, Ma Y, Wang H, Zhang J, Yuan J, Lin CP, Nowson C, MacGregor GA. School based education programme to reduce salt intake in children and their families (School-EduSalt): cluster randomised controlled trial. BMJ. 2015 Mar 18;350:h770. doi: 10.1136/bmj.h770. PMID 25788018
- [Derived] He FJ, Wu Y, Ma J, Feng X, Wang H, Zhang J, Lin CP, Yuan J, Ma Y, Yang Y, Yan LL, Jan S, Nowson C, Macgregor GA. A school-based education programme to reduce salt intake in children and their families (School-EduSalt): protocol of a cluster randomised controlled trial. BMJ Open. 2013 Jul 16;3(7):e003388. doi: 10.1136/bmjopen-2013-003388. Print 2013. PMID 23864214